CLINICAL TRIAL: NCT02925715
Title: Comparative Evaluation of Ultrasound Guided Supraclavicular and Infraclavicular Subclavian Venous Catheterizations in Adult Patients Undergoing Major Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Vikas Saini, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: INT/IEC/2015/321
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Compare Central Line Insertion of Subclavian Vein With Two Different Approaches Using Ultrasound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supraclavicular (Experimental): ultrasound guided central venous cannulation done by supraclavicular approach
  Interventions: Procedure: ultrasound guided central venous cannulation
- infraclavicular (Experimental): ultrasound guided central venous cannulation done by infraclavicular approach
  Interventions: Procedure: ultrasound guided central venous cannulation

INTERVENTIONS:
Procedure: ultrasound guided central venous cannulation — ultrasound is a medical device which is frequently used for safe venous punctures as you can visualise the structures.so, device ''ultrasound'' will be used for intervention ''central line insertion'' in subclavian vein. ultrasound guided cannulation of the subclavian vein was done by supraclavicular or infraclavicular approach after randomization into either of the two groups.In the supraclavicular approach the puncture site is above the clavicle while in the infraclavicular group the puncture site is below the clavicle. Central venous cannulation is done after identifying the vein on ultrasound and using standard seldinger technique with full asepsis.

SUMMARY:
Comparison of two techniques of central venous cannulation of subclavian vein using ultrasound was performed. ultrasound guided central venous cannulation is the standard practice today but its use in subclavian vein is technically challenging and not much literature is available. In this study 96 Patients were randomized into one of the groups and compared for various outcomes. The primary outcome studied was the time taken for procedure. Secondary objectives included comparison of total access time using both the techniques,comparison of first attempt success rate, comparison of the quality of needle visualization and the comparison of immediate (mechanical) and delayed complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults requiring central venous cannulation.

Exclusion Criteria:

* History of prior catheterization.
* Limited sites for access attempts (other catheters, pacemaker, prior surgery).
* Previous difficulties during catheterization such as more than three punctures at one site, two sites attempted or failure to gain access.
* Previous mechanical complications during catheterization.
* Patients with infection at puncture site and contralateral pneumothorax.
* Patients with trauma to clavicle and upper ribs, distorted anatomy of neck or clavicles.
* Cervical spine injury.
* Known vascular abnormality.
* Untreated coagulopathy such as International Normalization Ratio(INR) ≥ 2, activated partial thromboplastin time >1.5 of normal or platelets <50,000/mm3
* After 3 attempts at needle puncture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
puncture time of subclavian vein using ultrasound-guided supraclavicular or infraclavicular approach infraclavicular approaches in adults | 1 year
  will be measured in seconds

SECONDARY OUTCOMES:
total time taken for cannulation of veins using both the techniques. | 1 year
  measured in seconds
first attempt success rate | 1 year
  number of attempts taken will be measured
quality of needle visualisation | 1 year
  subjective visualisation of the needle on ultrasound will be noted as good or poor
immediate and delayed complications with the two approaches | 1 year